CLINICAL TRIAL: NCT07044089
Title: Comparison of Individualized PEEP Application Versus Fixed PEEP Application for Lung-Protective Ventilation in Patients Undergoing On-Pump Coronary Artery Bypass Grafting Surgery
Brief Title: Lung Protective Ventilation and Driving Pressure Guided PEEP Titration in CABG Surgery
Status: Recruiting | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zeynep AÇIK, Research Assistant Doctor, Kocaeli University
Other Study IDs: KAEK/05.b1.01
Record Dates: First submitted 2025-06-23; First posted 2025-06-29 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Peep Titration in Lung Protective Ventilation
Keywords: Lung Protective Ventilation; Fixed PEEP; Individualized PEEP

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fixed PEEP
- Indıvıdalızed PEEP

SUMMARY:
Our aim in this study is to compare fixed and individualized PEEP (driving pressure guided ) application for intraoperative lung protective ventilation in patients undergoing on-pump CABG surgery.

Researcher aimed to compare the effects of two different PEEP application methods on intraoperative hemodynamics, respiratory mechanics, and gas exchange, as well as postoperative extubation times, respiratory complications (atelectasis, need for non invasive mechanical ventilatıon, need for re-entubatıon) length of stay in the intensive care unit, and discharge times.

DETAILED DESCRIPTION:
The primary goal of the researchers: To compare the effects of fixed PEEP versus driving pressure guided individualized PEEP in lung protective mechanical ventilation during on-pump open heart surgery effect of PaO2/ FiO2 ratio end of surgery.

The secondary goals of the researchers: To compare intraoperative hemodynamics, lung compliance and airway pressures, extubation time and respiratory complications [development of atelectasis, need for noninvasive mechanical ventilation (high-flow nasal cannula or CPAP application), need for re-intubation], length of stay in the ICU and discharge times.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective on-pump coronary artery bypass graft surgery via median sternotomy
* Patients between the ages of 18 and 70
* ASA (American Society of Anesthesiologists) physical status classification II-III

Exclusion Criteria:

* Patients with an ejection fraction below 35%
* Patients who did not consent to participate in the study
* Patients undergoing emergency surgery
* Patients who are allergic to the anesthetic drugs used
* Patients who have undergone lung resection
* Those with a history of mechanical ventilation in the 2 months before surgery
* Patients who have undergone total circulatory arrest and deep hypothermia
* Patients with obstructive sleep apnea syndrome requiring long-term ventilation assistance
* Morbid obesity (Body Mass Index>35kg/m2)
* Patients with refractory hypoxemia (arterial oxygen saturation below 88% despite 100% oxygen inhalation)
* COPD (FEV1<70%)
* Patients with chronic renal failure (serum creatine>1.8 mg/dl)
* Anemia (Hg<10 gr/dl)
* Patients who have had an intraaortic balloon pump placed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo elective on-pump coronary artery bypass graft surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Effects on intraoperative oxygenation, hemodynamics, lung compliance and airway pressures | First one day
  Data will be recorded during surgery and the first 24 hours after extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Faculty of Medicine, Kocaeli, izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes